CLINICAL TRIAL: NCT03741725
Title: Pay-it-forward Gonorrhea and Chlamydia Testing Among Men Who Have Sex With Men in China: a Cluster Randomized Controlled Trial
Brief Title: Pay-it-forward RCT for Gonorrhea and Chlamydia Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Aging (NIA) (NIH); Southern Medical University, China (Other); London School of Hygiene and Tropical Medicine (Other); Social Entrepreneurship to Spur Health (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18-2142; 5P30AG034420-10 (NIH); R01AI114310 (NIH)
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-01

CONDITIONS: Gonorrhea Male; Chlamydia;M

STUDY DESIGN:
Intervention Model Description: 3-arm superiority randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pay-it-forward (Experimental): First, participants will be provided a brief introduction to gonorrhea and chlamydia testing. Then, participants will be offered a gift of free gonorrhea and chlamydia testing made available by donations from previous testers, and asked whether they would like to donate money (pay-it-forward) for future men to receive the same option.
  Interventions: Other: Pay-it-forward
- Pay-what-you-want (Experimental): First, participants will be provided a brief introduction to gonorrhea and chlamydia testing. Then, participants will be offered gonorrhoea and chlamydia testing and told that they can decide and pay any desired amount after receiving the test.
  Interventions: Other: Pay-what-you-want
- Standard of care (No Intervention): First, participants will be provided a brief introduction to gonorrhea and chlamydia testing. Then, participants will be offered gonorrhoea and chlamydia testing at the standard patient price.

INTERVENTIONS:
Other: Pay-it-forward — Participants will be offered a gift of free gonorrhea and chlamydia testing made available by donations from previous testers, and asked whether they would like to donate money (pay-it-forward) for future men to receive the same option.
  Arms: Pay-it-forward
Other: Pay-what-you-want — Participants will be offered gonorrhoea and chlamydia testing and told that they can decide and pay any desired amount after receiving the test.
  Arms: Pay-what-you-want

SUMMARY:
This is a randomized controlled trial which will evaluate dual gonorrhea/chlamydia test uptake and other outcomes in men who have sex with men (MSM) in three trial arms - 1) a pay-it-forward testing arm, 2) a pay-what-you-want testing arm, and 3) standard of care arm.

DETAILED DESCRIPTION:
At both of the program sites, MSM partaking in HIV and syphilis testing will be offered dual gonorrhea/chlamydia testing. First, all men will be provided a brief (5 minute) introduction to gonorrhea and chlamydia testing using a pamphlet. Program organizers will then explain the pay-it-forward program to each man separately. Briefly, men will be told that the hospital list price of gonorrhea and chlamydia testing was 150 RMB ($24 USD), but previous men attending the clinic had donated money to cover the cost of his test. Thus, each man could receive a free gonorrhea and chlamydia test, then decide whether to donate money (pay-it-forward) for future men to receive the same option. Men will be assured that donating is completely optional and advised to pay any amount that is feasible for them. Each man's gonorrhea and chlamydia test fees will be covered by a combination of the initial funding pool from the program organizers and the donations from previous participants. Men will also be shown a postcard with a message written by a previous pay-it-forward contributor. Messages will contain information encouraging men to be tested/slogans to promote sexual health and testing (i.e. taking ownership of their health). They will be told that they could also write a postcard message for a future participant.

Men will then decide whether or not to receive combined urine gonorrhea/chlamydia testing. Program organizers will inform participants of their test results via WeChat. Patients with positive test results will be counseled and directed to the WeChat page of designated hospitals where they could make an appointment to receive treatment and follow-up.

ELIGIBILITY:
Inclusion criteria:

* born biologically male
* age 16 years or older
* report previous anal sex with another man
* willing to provide mobile phone number for results notification

Exclusion criteria:

* tested for both gonorrhoea and chlamydia in the past 12 months with no high-risk sexual behavior following testing
* previous participation in pay-it-forward program

Ages: 16 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 301 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tucker, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- China (3):
  - Southern Medical University, Guangzhou, Guangdong
  - Zhitong Guangzhou LGBT Center, Guangzhou, Guangdong
  - BlueD Danlan Happy Testing Office, Beijing

REFERENCES:
- [Background] Li KT, Tang W, Wu D, Huang W, Wu F, Lee A, Feng H, Pan SW, Han L, Mak V, Yang L, Tucker JD. Pay-it-forward strategy to enhance uptake of dual gonorrhea and chlamydia testing among men who have sex with men in China: a pragmatic, quasi-experimental study. Lancet Infect Dis. 2019 Jan;19(1):76-82. doi: 10.1016/S1473-3099(18)30556-5. PMID 30587296
- [Background] Zhang TP, Liu C, Han L, Tang W, Mao J, Wong T, Zhang Y, Tang S, Yang B, Wei C, Tucker JD. Community engagement in sexual health and uptake of HIV testing and syphilis testing among MSM in China: a cross-sectional online survey. J Int AIDS Soc. 2017 Apr 3;20(1):21372. doi: 10.7448/IAS.20.01.21372. PMID 28406270
- [Derived] Yang F, Zhang TP, Tang W, Ong JJ, Alexander M, Forastiere L, Kumar N, Li KT, Zou F, Yang L, Mi G, Wang Y, Huang W, Lee A, Zhu W, Luo D, Vickerman P, Wu D, Yang B, Christakis NA, Tucker JD. Pay-it-forward gonorrhoea and chlamydia testing among men who have sex with men in China: a randomised controlled trial. Lancet Infect Dis. 2020 Aug;20(8):976-982. doi: 10.1016/S1473-3099(20)30172-9. Epub 2020 Apr 28. PMID 32530426
- [Derived] Zhang TP, Yang F, Tang W, Alexander M, Forastiere L, Kumar N, Li K, Zou F, Yang L, Mi G, Wang Y, Huang W, Lee A, Zhu W, Vickerman P, Wu D, Yang B, Christakis NA, Tucker JD. Pay-it-forward gonorrhea and chlamydia testing among men who have sex with men in China: a study protocol for a three-arm cluster randomized controlled trial. Infect Dis Poverty. 2019 Aug 16;8(1):76. doi: 10.1186/s40249-019-0581-1. PMID 31426869

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: cluster of participants
Groups:
- Pay-it-forward: First, participants were provided a brief introduction to gonorrhea and chlamydia testing. Then, participants were offered a gift of free gonorrhea and chlamydia testing made available by donations from previous testers, and asked whether they would like to donate money (pay-it-forward) for future men to receive the same option.
  Pay-it-forward: Participants were offered a gift of free gonorrhea and chlamydia testing made available by donations from previous testers, and asked whether they would like to donate money (pay-it-forward) for future men to receive the same option.
- Pay-what-you-want: First, participants were provided a brief introduction to gonorrhea and chlamydia testing. Then, participants were offered gonorrhoea and chlamydia testing and told that they could decide and pay any desired amount after receiving the test.
  Pay-what-you-want: Participants were offered gonorrhoea and chlamydia testing and told that they could decide and pay any desired amount after receiving the test.
- Standard of Care: First, participants were provided a brief introduction to gonorrhea and chlamydia testing. Then, participants were offered gonorrhoea and chlamydia testing at the standard patient price.
Period: Overall Study
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Started | 101; 10 cluster of participants | 100; 10 cluster of participants | 100; 10 cluster of participants
Completed | 101; 10 cluster of participants | 100; 10 cluster of participants | 100; 10 cluster of participants
Not Completed | 0; 0 cluster of participants | 0; 0 cluster of participants | 0; 0 cluster of participants

BASELINE CHARACTERISTICS:
Population: Each arm had ten clusters of participants.
Groups:
- Pay-it-forward: Men in pay-it-forward were told that the standard price of the gonorrhea and chlamydia testing was 150RMB ($22US), and that previous participants who cared about them donated toward testing fees. Thus, men in the pay-it-forward arm received a free test, and then decided whether, and if so how much to donate toward future testing for others. Participants were shown postcards and told that testing and donating were voluntary.
- Pay-what-you-want: After being introduced to the testing and the study, men in the pay-what-you-want arm were told that the standard price of gonorrhea and chlamydia testing was 150RMB ($22US), and that they would receive free testing and then decide the amount that they would like to pay for their own test.
- Standard-of-care: Men in the standard of care arm received the same introduction to gonorrhea and chlamydia testing as the men in the other two arms. They were then told that the standard price of gonorrhea and chlamydia testing was 150RMB (US$22) and they had to pay the full amount for the their testing.
- Total: Total of all reporting groups
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard-of-care | Total
Number analyzed (Participants) | 101 | 100 | 100 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them.
  years
    number analyzed (Participants) | 98 | 93 | 97 | 288
    (all) | 28.6 (7.8) | 26.6 (5.6) | 29.1 (7.5) | 28.1 (7.1)
Age, Customized [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them.
  Participants
    number analyzed (Participants) | 98 | 93 | 97 | 288
    <= 30 years | 66 | 74 | 66 | 206
    >30 years | 32 | 19 | 31 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 101 | 100 | 100 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 100 | 100 | 301
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 101 | 100 | 100 | 301
Marital status [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them.
  Participants
    number analyzed (Participants) | 98 | 93 | 97 | 288
    Never married | 87 | 84 | 81 | 252
    Other (engaged, married, divorced or separated) | 11 | 9 | 16 | 36
Highest education completed [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them.
  Participants
    number analyzed (Participants) | 98 | 93 | 97 | 288
    Middle school or below | 5 | 5 | 6 | 16
    High/vocational school | 8 | 9 | 10 | 27
    College or above | 85 | 79 | 81 | 245
Annual income (USD) [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them.
  Participants
    number analyzed (Participants) | 98 | 93 | 97 | 288
    <2,680 | 11 | 13 | 9 | 33
    2,681- 5,360 | 7 | 9 | 10 | 26
    5,361- 8,934 | 17 | 15 | 11 | 43
    8,935- 14,294 | 23 | 23 | 30 | 76
    >14,294 | 40 | 33 | 37 | 110
Number of sex partners in the past three months, Categorical [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them. Two additional participants in pay-it-forward, two in pay-what-you-want, and six in standard-of-care did not respond to this question.
  Participants
    number analyzed (Participants) | 96 | 91 | 91 | 278
    0-1 | 47 | 47 | 42 | 136
    Multiple | 49 | 44 | 49 | 142
Had anal sex in the past three months [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them. One additional person in standard-of-care did not respond to this specific survey question.
  Participants
    number analyzed (Participants) | 98 | 93 | 96 | 287
    Yes | 84 | 73 | 77 | 234
    No | 14 | 20 | 19 | 53
Condom use frequency during anal sex in the past three months [Count of Participants; unit: Participants] — Population: Only participants who reported having had anal sex in the past three months were asked this question about condom use during anal sex.
  Participants
    number analyzed (Participants) | 84 | 73 | 77 | 234
    Non-use | 5 | 5 | 4 | 14
    Sometimes | 6 | 9 | 9 | 24
    Often | 21 | 24 | 24 | 69
    Always | 52 | 35 | 40 | 127
HIV testing frequency in the past two years [Count of Participants; unit: Participants] — Population: 3 in pay-it-forward arm, 7 in pay-what-you-want arm, and 3 in standard-of-care arm did not complete or submit their survey questionnaires. Hence, demographic and behavioral information is lacking for them. One additional participant in the standard-of-care arm did not respond to this specific survey question.
  Participants
    number analyzed (Participants) | 98 | 93 | 96 | 287
    Never tested | 6 | 14 | 6 | 26
    < once every two years | 15 | 9 | 9 | 33
    Once a year | 23 | 16 | 24 | 63
    Every six months | 26 | 24 | 26 | 76
    Every three months | 21 | 25 | 27 | 73
    Monthly | 7 | 5 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received the Dual Gonorrhea/Chlamydia Testing
Description: Dual gonorrhea/chlamydia test uptake as assessed by administrative records in each arm.
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard-of-care
Number analyzed (Participants) | 101 | 100 | 100
Participants | 57 | 46 | 18

2. Secondary Outcome: Number of Participants Tested Positive for Gonorrhea
Description: The number of men who tested positive for gonorrhea through this study. Samples were collected either from urine or rectum.
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Population: Overall Number of Participants Analyzed include the participants who received the Dual Gonorrhea/Chlamydia Testing
Measure: Count of Participants; unit: Participants
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 57 | 46 | 18
Participants | 1 | 2 | 2

3. Secondary Outcome: Number of Participants Tested Positive for Chlamydia
Description: The is the number of men who tested positive for chlamydia through this study
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Population: Overall Number of Participants Analyzed include the participants who received the Dual Gonorrhea/Chlamydia Testing
Measure: Count of Participants; unit: Participants
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 57 | 46 | 18
Participants | 8 | 8 | 3

4. Secondary Outcome: Cost Per Test
Description: Cost per test, defined as the cost associated with respective interventions (development, start-up, implementation, intervention) per individual who reported testing for gonorrhea and chlamydia following the intervention; economic test and financial cost are reported separately.
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 101 | 100 | 100
USD
  Using economic cost | 11.24 (1.64) | 9.67 (1.46) | 6.12 (1.12)
  Using financial cost | 6.52 (1.48) | 6.56 (1.26) | 1.46 (0.62)

5. Secondary Outcome: Cost Per Diagnosis
Description: Cost per diagnosis, defined as the cost associated with respective interventions (development, start-up, implementation, intervention) per individual who tested positive for gonorrhea and/or chlamydia following the intervention. Cost using economic cost and financial cost were respectively reported.
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Measure: Mean (Standard Error); unit: USD
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 101 | 100 | 100
USD
  Using economic cost | 11.24 (1.66) | 9.67 (1.45) | 6.12 (1.13)
  Using financial cost | 6.52 (1.47) | 6.56 (1.29) | 1.46 (0.62)

6. Secondary Outcome: Number of Participants Reporting Community Engagement Activities
Description: Number of participants who reported yes/no to specific questions on the awareness of and/or participation in MSM-related causes, organizations, or community events
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Population: Those are participants who filled out this questionnaire among those who participated in the study. In total, 3 participants did not respond in Pay-it-for-ward, 7 in Pay-what-you-want, and 3 in Standard of Care.
Measure: Count of Participants; unit: Participants
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 98 | 93 | 97
Participants
  Have you ever participated in online forums or dis: number analyzed (Participants) | 95 | 92 | 90
  Have you ever participated in online forums or dis: Yes | 78 | 64 | 61
  Have you ever participated in online forums or dis: No | 17 | 28 | 29
  Are you aware of any ongoing MSM-related community: number analyzed (Participants) | 93 | 92 | 89
  Are you aware of any ongoing MSM-related community: Yes | 48 | 30 | 37
  Are you aware of any ongoing MSM-related community: No | 45 | 62 | 52
  Have you ever encouraged someone to use MSM-relate: number analyzed (Participants) | 93 | 92 | 88
  Have you ever encouraged someone to use MSM-relate: Yes | 77 | 72 | 70
  Have you ever encouraged someone to use MSM-relate: No | 16 | 20 | 18
  Have you ever attended MSM-related community event: number analyzed (Participants) | 94 | 92 | 92
  Have you ever attended MSM-related community event: Yes | 31 | 23 | 23
  Have you ever attended MSM-related community event: No | 63 | 69 | 69
  Have you ever donated to MSM-related causes, event: number analyzed (Participants) | 96 | 92 | 94
  Have you ever donated to MSM-related causes, event: Yes | 41 | 30 | 23
  Have you ever donated to MSM-related causes, event: No | 55 | 62 | 71
  Have you ever volunteered for MSM-related causes: number analyzed (Participants) | 93 | 91 | 90
  Have you ever volunteered for MSM-related causes: Yes | 19 | 13 | 14
  Have you ever volunteered for MSM-related causes: No | 74 | 78 | 76

7. Secondary Outcome: Community Connectedness Scale Scores
Description: Community connectedness scales include six statements and Likert scale response ranging from 1= Strongly disagree, 2= Agree, 3= Disagree, and 4= Strongly agree.
  For each scale item, the range spans across 1 to 4, with higher score indicating more agreement with the statement and potentially higher community connectedness.
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Population: Some participants declined to answer certain questions. Hence, the number analyzed in some rows is different from the overall number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 98 | 93 | 97
score on a scale
  You feel that you are a part of the MSM community.: number analyzed (Participants) | 98 | 92 | 93
  You feel that you are a part of the MSM community. | 3.32 (0.74) | 3.05 (0.72) | 3.10 (0.63)
  Participating in MSM community is a positive thing: number analyzed (Participants) | 98 | 92 | 93
  Participating in MSM community is a positive thing | 3.16 (0.77) | 3.00 (0.73) | 3.00 (0.59)
  You are proud of the MSM community: number analyzed (Participants) | 97 | 92 | 90
  You are proud of the MSM community | 2.75 (0.87) | 2.71 (0.73) | 2.78 (0.78)
  Important for you to advocate for the community: number analyzed (Participants) | 98 | 92 | 92
  Important for you to advocate for the community | 3.24 (0.67) | 3.23 (0.59) | 3.10 (0.70)
  If you all work together, problems will be solved: number analyzed (Participants) | 97 | 91 | 92
  If you all work together, problems will be solved | 2.92 (0.83) | 2.86 (0.69) | 2.88 (0.69)
  Any problems faced by the MSM are also yours: number analyzed (Participants) | 97 | 91 | 92
  Any problems faced by the MSM are also yours | 3.22 (0.60) | 3.13 (0.62) | 3.02 (0.63)

8. Secondary Outcome: Social Cohesion Scale Scores
Description: Social cohesion is a scale made of seven statements and Likert response to them ranging from 1= strongly disagree, 2 = disagree, 3 = agree, and 4= strongly agree. Those questions asked about the feelings of being able to depend on a larger MSM community (i.e., tongzhi circle, gay online networks or groups).
  For each item, the range spans across 1 to 4. For items 1 to 5, the higher score, the more agreement with the statement and potentially the higher social cohesion. Item 6 and 7 are reversely scored, meaning that the higher the score, the lower social cohesion potentially.
Time Frame: During enrollment visit, an approximate total of 1.5 hours
Population: Some participants chose to decline certain questions, which resulted in numbers analyzed in some rows being different from the overall number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard of Care
Number analyzed (Participants) | 98 | 93 | 97
score on a scale
  You can count on other MSM to lend money: number analyzed (Participants) | 98 | 92 | 91
  You can count on other MSM to lend money | 2.52 (0.84) | 2.57 (0.76) | 2.64 (0.72)
  You can count on other MSM to talk about problems: number analyzed (Participants) | 98 | 92 | 93
  You can count on other MSM to talk about problems | 2.98 (0.69) | 2.86 (0.75) | 2.98 (0.53)
  You can count on other MSM if you need a place: number analyzed (Participants) | 98 | 92 | 93
  You can count on other MSM if you need a place | 2.71 (0.81) | 2.73 (0.76) | 2.73 (0.71)
  MSM you socialize with is an integrated group: number analyzed (Participants) | 98 | 92 | 92
  MSM you socialize with is an integrated group | 2.63 (0.71) | 2.68 (0.73) | 2.66 (0.68)
  You can trust the majority of the MSM you know.: number analyzed (Participants) | 98 | 92 | 93
  You can trust the majority of the MSM you know. | 2.74 (0.71) | 2.59 (0.71) | 2.61 (0.66)
  MSM in your group only worry about themselves: number analyzed (Participants) | 98 | 92 | 92
  MSM in your group only worry about themselves | 2.48 (0.71) | 2.54 (0.76) | 2.47 (0.67)
  MSM you socialize with are always arguing: number analyzed (Participants) | 98 | 92 | 93
  MSM you socialize with are always arguing | 2.31 (0.69) | 2.18 (0.77) | 2.26 (0.62)

ADVERSE EVENTS:
Time Frame: Time frame was during one study visit on the day of participation.
Arm/Group | Pay-it-forward | Pay-what-you-want | Standard-of-care
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03741725/Prot_SAP_000.pdf